CLINICAL TRIAL: NCT06466135
Title: Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of WAL0921 in Patients With Glomerular Kidney Diseases and Proteinuria
Brief Title: Study of WAL0921 in Patients With Glomerular Kidney Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Walden Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WAL0921-02
Record Dates: First submitted 2024-06-12; First posted 2024-06-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Nephropathies; Primary Focal Segmental Glomerulosclerosis; Minimal Change Disease; Primary Immunoglobulin A Nephropathy; Primary Membranous Nephropathy
Keywords: DN; FSGS; TR-MCD; IgAN; PMN
MeSH Terms: conditions — Diabetic Nephropathies; Nephrosis, Lipoid; Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WAL0921 (Experimental): Intravenous infusion of investigational drug WAL0921
  Interventions: Drug: WAL0921
- Placebo (Placebo Comparator): Intravenous infusion of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WAL0921 — Investigational drug WAL0921 Participants receive an intravenous infusion of WAL0921 investigational drug once every 2 weeks for 7 total infusions.
  Arms: WAL0921
Drug: Placebo — Placebo product Participants receive an intravenous infusion of placebo once every 2 weeks for 7 total infusions.
  Arms: Placebo

SUMMARY:
This is an adaptive prospective, multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety, efficacy, pharmacokinetics, and pharmacodynamics of WAL0921 in subjects with glomerular kidney disease and proteinuria, including diabetic nephropathy and rare glomerular kidney diseases (primary focal segmental glomerulosclerosis [FSGS], treatment-resistant minimal change disease [TR MCD], primary immunoglobulin A nephropathy [IgAN], and primary membranous nephropathy [PMN]). Subjects in this study will be randomized to receive the investigational drug WAL0921 or placebo as an intravenous infusion once every 2 weeks for 7 total infusions. All subjects will be followed for 24 weeks after their last infusion.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-75 years
* Diagnosis of one of the following glomerular kidney diseases: diabetic nephropathy; primary focal segmental glomerulosclerosis; treatment resistant-minimal change disease; primary IgA nephropathy; primary membranous nephropathy
* eGFR greater than or equal to 30 mL/min/1.73 m2

Exclusion Criteria:

* Currently pregnant or planning to become pregnant
* History of organ transplantation
* History of alcohol or substance use disorder
* Acute dialysis or acute kidney injury within 6 months of Screening
* Any prior or current medical condition that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Baseline to Week 36

SECONDARY OUTCOMES:
Change in albuminuria | Baseline up to Week 24
  Percent change in urine albumin-creatinine ratio (UACR)
Change in proteinuria | Baseline up to Week 24
  Percent change in urine protein-creatinine ratio (UPCR)
Change in estimated glomerular filtration rate | Baseline up to Week 24
  Percent change in estimated glomerular filtration rate (eGFR)
Change in rate of change in eGFR | Baseline up to Week 24
  Slope of eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blair, MD, Study Director — Walden Biosciences
Locations (9):
- United States (2):
  - Colorado Kidney and Vascular Care, Denver, Colorado
  - D & H Tamarac Research Center, Tamarac, Florida
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Western Health Sunshine Hospital, St Albans, Victoria
- United Kingdom (5):
  - Royal Derby Hospital, Derby
  - College of Life Sciences, University of Leicester, Leicester
  - Barts Health NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Salford Royal NHS Foundation Trust, Salford